CLINICAL TRIAL: NCT03001960
Title: Dual AntiPlatelet Therapies for Prevention of Periinterventional Embolic Events in Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: Dual AntiPlatelet Therapies for Prevention of Periinterventional Embolic Events in TAVI
Acronym: DAPT-TAVI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. Dr. Jochen Fiebach, Center for Stroke Research Berlin (CSB), Charité - Universitaetsmedizin Berlin (Unknown)
Responsible Party: Principal Investigator, Alexander Lauten, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPT-TAVI 01
Record Dates: First submitted 2016-12-18; First posted 2016-12-23 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement; Intracranial Embolism
MeSH Terms: conditions — Aortic Valve Stenosis; Intracranial Embolism | interventions — Argininosuccinate Synthase; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1- PREloading BEFORE TAVI (Experimental): * Aspirin 100 mg loading orally 6-12 hours before TAVI and
  * Clopidogrel 600mg loading 6-12 before TAVI followed by maintenance dose of 100mg aspirin and 75mg clopidogrel per day
  Interventions: Drug: Preloading before TAVI
- Group 2 - POSTLoading AFTER TAVI (Experimental): * Aspirin 100 mg loading orally 6-12 hours after TAVI and
  * Clopidogrel 600mg loading 6-12 hours after TAVI followed by maintenance dose of 100mg aspirin and 75mg clopidogrel per day
  Interventions: Drug: Postloading after TAVI

INTERVENTIONS:
Drug: Preloading before TAVI — Preloading with Aspirin and Clopidogrel before TAVI
  Other Names: ASS, Plavix
  Arms: Group 1- PREloading BEFORE TAVI
Drug: Postloading after TAVI — Postloading with Aspirin and Clopidogrel after TAVI
  Other Names: ASS, Plavix
  Arms: Group 2 - POSTLoading AFTER TAVI

SUMMARY:
TAVI is increasingly adopted as standard treatment for many subgroups of patients with aortic stenosis. However, due to a lack of data there is yet no TAVI-specific guidance regarding the optimum periinterventional drug regimen.

The study evaluates the effect of dual antiplatelet pretreatment on periinterventional embolic cerebral lesions and bleeding complications in patients undergoing transfemoral aortic valve implantation (TF-TAVI).

DETAILED DESCRIPTION:
Patients undergoing TAVI bear a high risk of ischaemic stroke, which is an independent predictor of mortality1. Dual antiplatelet therapy (DAPT) is recommended by current guidelines without clear specifications on the time of initiation of treatment due to a lack of data. While some centers initiate DAPT with aspirin and clopidogrel prior to TAVI to reduce the rate of periinterventional embolic events, others start these medications after the procedure.Data on antithrombotic therapy during TAVI are scarce and no randomized evaluation has been performed to demonstrate what the best strategy is during the procedure.

Therefore, the objective of this clinical trial is to assess the efficacy of pre- versus postoperative dual antiplatelet loading with Aspirin and Clopidogrel on volume of periinterventional cerebral ischemic lesions as quantified by diffusion weight MRI (DW-MRI) and neurocognitive function in patients undergoing transfemoral aortic valve replacement. The statistical trial design assumes superiority of preloading with DAPT regarding the primary endpoint.

ELIGIBILITY:
Inclusion criteria:

* Patients >18 years and <90 years
* Patients undergoing TF-TAVI for severe aortic stenosis (combined with aortic regurgitation)
* Informed consent

Exclusion criteria:

* TIA/Stroke within last 90 days
* Aortic valve-in-valve procedures
* TAVI for treatment of isolated aortic regurgitation
* known significant carotid stenosis (>70%)
* Prior myocardial infarction or revascularization with PCI or CABG within past 3 months
* Clopidogrel and/ or Aspirin within past 7 days
* any other indication for (dual) antiplatelet therapy
* Contraindication to MRI (MRI conditional pacemakers accepted!)
* participation in another interventional trial
* cardiogenic shock (positive shock index OR need for catecholamine support OR systolic bloodpressure < 90 mmHg) or need for pre-hospital intubation
* cardiac arrest <90 days prior to randomization
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Total volume of new cerebral lesions on MRI after TAVI versus Baseline | Total volume of new cerebral lesions on MRI, 24-72h after TAV versus Baseline

SECONDARY OUTCOMES:
New lesion volume of cerebral embolization in patients treated with ASS and Clopidogrel before versus after TAVI | 24-72h post TAVI versus baseline
  Total new lesion volume is defined as the sum volume of all new cerebral ischemic lesions on the post-procedural MRI relative to the pre-TAVR cerebral MRI scan (on diffusion weighted and FLAIR MRI images).
location of new cerebral lesions early AFTER TAVI | 24-72h after TAVI
  To evaluate cerebral embolisation, which is not procedure related, cerebral embolisation on MRI will be before TAVI versus the post-TAVI MRI scan
extent of new cerebral lesions early AFTER TAVI | 24-72h after TAVI
  To evaluate cerebral embolisation, which is not procedure related, cerebral embolisation on MRI will be before TAVI versus the post-TAVI MRI scan
Assessment of different neurocognitive tests before and after TAVI procedure | 24-72 h after TAVI
  To evaluate neurologic function with a battery of neurocognitive tests and to correlate these findings to cerebral MRI scans
Extent of clinically apparent non-cerebral emboli after TAVI | 24-72 h after TAVI
  To describe extent and localization of non-cerebral embolisation (e.g. pulmonary embolism, limb ischaemia...)
localization of clinically apparent non-cerebral emboli after TAVI | 24-72 h after TAVI
  To describe extent and localization of non-cerebral embolisation (e.g. pulmonary embolism, limb ischaemia...)
Evaluation of possible changes in quality of life after TAVI with EQ-5D questionnaire sum score. | 24-72 h after TAVI

REFERENCES:
- [Background] Holmes DR Jr, Brennan JM, Rumsfeld JS, Dai D, O'Brien SM, Vemulapalli S, Edwards FH, Carroll J, Shahian D, Grover F, Tuzcu EM, Peterson ED, Brindis RG, Mack MJ; STS/ACC TVT Registry. Clinical outcomes at 1 year following transcatheter aortic valve replacement. JAMA. 2015 Mar 10;313(10):1019-28. doi: 10.1001/jama.2015.1474. PMID 25756438
- [Background] Osnabrugge RL, Mylotte D, Head SJ, Van Mieghem NM, Nkomo VT, LeReun CM, Bogers AJ, Piazza N, Kappetein AP. Aortic stenosis in the elderly: disease prevalence and number of candidates for transcatheter aortic valve replacement: a meta-analysis and modeling study. J Am Coll Cardiol. 2013 Sep 10;62(11):1002-12. doi: 10.1016/j.jacc.2013.05.015. Epub 2013 May 30. PMID 23727214